CLINICAL TRIAL: NCT03506477
Title: A Double-blinded, Placebo-controlled Study to Evaluate the Tolerability and Efficacy of Enstilar® (Calcipotriene and Betamethasone Dipropionate) Foam in the Treatment of Chronic Plaque Psoriasis in Patients With Skin of Color
Brief Title: Enstilar® Foam in the Treatment of Chronic Plaque Psoriasis in Patients With Skin of Color
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Icahn School of Medicine at Mount Sinai (Other)
Responsible Party: Principal Investigator, Andrew Alexis, MD, Chair, Department of Dermatology, Icahn School of Medicine at Mount Sinai
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: GCO 17-2468; HSM# 17-05032 (Other: Icahn School of Medicine at Mount Sinai)
Record Dates: First submitted 2018-04-17; First posted 2018-04-24 (Actual); Results first posted 2021-01-20 (Actual); Last update posted 2021-01-20 (Actual); Status verified 2020-09

CONDITIONS: Plaque Psoriasis; Psoriasis
Keywords: skin of color; psoriasis; Enstilar; skin diseases
MeSH Terms: conditions — Psoriasis; Skin Diseases | interventions — betamethasone dipropionate, calcipotriol drug combination

STUDY DESIGN:
Intervention Model Description: 4:1 Enstilar(R): placebo from baseline to week 4, then open-label Enstilar from weeks 4 to 8.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Double-blind, vehicle-controlled from week 0 to 4
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Enstilar® foam (Experimental): Enstilar® foam - a combination of calcipotriene and betamethasone dipropionate 0.005%/0.064%.
  Interventions: Drug: Enstilar® foam
- Vehicle foam (Placebo Comparator): does not contain the active ingredient
  Interventions: Drug: Vehicle foam

INTERVENTIONS:
Drug: Enstilar® foam — for 4 weeks
  Other Names: Enstilar 0.005%-0.064% Topical Foam
  Arms: Enstilar® foam
Drug: Vehicle foam — for 4 weeks
  Arms: Vehicle foam

SUMMARY:
This will be a single-center, randomized, double-blinded, vehicle-controlled clinical study to determine the efficacy of Enstilar® foam, a combination of calcipotriene and betamethasone dipropionate 0.005%/0.064%, in the treatment of psoriasis vulgaris in skin of color (FST IV-VI). This study will also evaluate the degree of erythema versus hyperpigmentation in psoriasis plaques in skin of color (and its change with Enstilar ® treatment) as well as the effect of Enstilar ® on post-inflammatory hyperpigmentation and quality of life.

DETAILED DESCRIPTION:
Psoriasis is a chronic inflammatory disorder primarily affecting the skin and joints. This condition occurs in different ethnic groups worldwide with varying prevalence.

There are notable differences in psoriasis presentation in skin of color groups. Black patients with psoriasis tend to have less erythema, increased risk of pigmentation, thicker plaques, more scaling, and greater body involvement as compared to white patients. The resolution of psoriasis lesions in darker skin types is associated with a higher rate of dyspigmentation (both hyper- and hypo-pigmentation), which may be more bothersome to patients than the psoriasis itself. Further, several studies have shown that psoriasis is associated with greater psychological impact and worse quality of life in non-whites with psoriasis compared to whites.

Unique issues in skin of color populations make studies dedicated to darker skin types essential for the treatment of psoriasis in these populations. This study will evaluate the efficacy of Enstilar® foam, a combination of calcipotriene and betamethasone dipropionate 0.005%/0.064%, in the treatment of psoriasis vulgaris in darker skin types. This study will also evaluate the degree of erythema versus hyperpigmentation in psoriasis plaques as well as the effect of Enstilar ® on post-inflammatory hyperpigmentation and quality of life in skin of color.

ELIGIBILITY:
Inclusion Criteria:

* Provide written, signed and dated informed consent prior to initiating any study-related activities.
* Male or female >18 years of age at the time of screening
* Fitzpatrick Skin phototype IV-VI, non-white race/ethnicity, including but not limited to - --African Americans, Asians, Pacific Islanders and Hispanics.
* Clinical diagnosis of chronic plaque-type psoriasis of the body
* Plaque psoriasis with ≥2% Body Surface Area (BSA) involvement (may include scalp involvement), PASI Score ≥ 2, IGA mod 2011 score of 2 or greater (based on scale of 0-4)
* Females of childbearing potential (FCBP) must have a negative pregnancy test at Screening and Baseline. While using investigational product and for at least 28 days after last application of investigational product, FCBP who engage in activity in which conception is possible must use one of the approved contraceptive options d
* Must be in general good health as judged by the Investigator, based on medical history and physical examination.

Exclusion Criteria:

* Form of diagnosed psoriasis other than chronic plaque psoriasis (i.e. guttate, erythrodermic, pustular)
* Diagnosis of other active, ongoing skin diseases or skin infections that may interfere with examination of psoriasis lesions
* Ongoing use of other psoriasis treatment including but not limited to topical or systemic corticosteroids, other topical medications (i.e. coal tar), oral or biologic medications for the treatment of psoriasis, and UV therapy. The following washout periods will be required: 2 weeks for topical therapy; 2 weeks for phototherapy; 12 weeks for biologic or targeted therapies; 4 weeks for other systemic therapies
* Use of oral estrogen therapy, excluding oral contraceptive pills
* Women who are pregnant, nursing, or of child-bearing potential who are unwilling to use appropriate method(s) of contraception.
* Patients unwilling to limit exposure to UV light
* Current significant medical problems that, in the discretion of the investigator, would put the patient at significant risk
* Patients with disorders of calcium metabolism and/or hypercalcemia
* Use of any investigational drug within 4 weeks prior to randomization, or 5 pharmacokinetic/pharmacodynamics half-lives, if known (whichever is longer)
* History of allergy to any component of the IP

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2018-05-21 (Actual); Primary Completion 2019-09-25 (Actual); Study Completion 2019-09-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Alexis, MD, MPH, Principal Investigator — Icahn School of Medicine at Mount Sinai
Locations (1):
- Mount Sinai West, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
With Leo, Pharma.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were recruited from the dermatology faculty practice and resident clinics in the Mount Sinai Health System from May 2018 through July 2019
Groups:
- Enstilar® Foam: Enstilar® foam x 4 weeks - a combination of calcipotriene and betamethasone dipropionate 0.005%/0.064%.
- Vehicle Foam: Vehicle foam: for 4 weeks - does not contain the active ingredient
Period: Overall Study
Arm/Group | Enstilar® Foam | Vehicle Foam
Started | 20 | 5
Completed | 19 | 5
Not Completed | 1 | 0
Not completed — Withdrawal by Subject | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Enstilar® Foam | Vehicle Foam | Total
Number analyzed (Participants) | 20 | 5 | 25
Age, Continuous [Mean (Standard Deviation); unit: years] | 49.6 (14.8) | 63.0 (8.9) | 50.3 (13.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 1 | 9
  Male | 12 | 4 | 16
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 7 | 2 | 9
  Not Hispanic or Latino | 13 | 3 | 16
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 2 | 1 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 1
  Black or African American | 12 | 1 | 13
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 6 | 2 | 8
IGA mod 2011 [Mean (Standard Deviation); unit: units on a scale] — Investigator's Global Assessment (2011 modified version ) (IGA mod 2011) is a five-category scale indicating the physician's overall assessment of psoriasis severity, by induration, erythema, and scaling, evaluated with categories of "0 = clear," "1 = almost clear," "2 = mild," "3 = moderate," or "4 = severe."
  units on a scale | 2.75 (0.54) | 2.8 (0.4) | 2.76 (0.51)
Scalp Investigator Global Assessment (ScIGA) [Mean (Standard Deviation); unit: units on a scale] — ScIGA ranges from 0 (clear) to 4 (severe). Population: Data only for those participants with scalp disease at baseline
  units on a scale
    number analyzed (Participants) | 12 | 4 | 16
    (all) | 2.25 (0.60) | 2.75 (0.83) | 2.38 (0.70)
Patient's Global Assessment of disease severity (PaGA) [Mean (Standard Deviation); unit: units on a scale] — PaGA have 5 distinct options ranging from (0) "Clear" to (4) "Severe."
  units on a scale | 3 (0.8) | 3.6 (0.49) | 3.16 (0.78)

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients Who Achieved Treatment Success
Description: Number of patients at week 4 who achieved treatment success according to Investigator's Global Assessment (IGA mod 2011) of the entire body including scalp. IGA ranges from 0 (clear) to 4 (severe). Treatment success is defined as IGA of clear (0) or almost clear (1) for patients with ≥ moderate disease at baseline or IGA of clear (0) for patients with mild disease at baseline.
Time Frame: Week 4
Measure: Count of Participants; unit: Participants
Arm/Group | Enstilar® Foam | Vehicle Foam
Number analyzed (Participants) | 19 | 5
Participants | 4 | 0

2. Secondary Outcome: Number of Participants With Achieving Targeted Psoriasis Area and Severity Index (PASI)
Description: Number of patients achieving ≥50% improvement and/or ≥75% improvement in PASI at weeks 4 and 8 . PASI combines the assessment of the severity of lesions and the area affected into a single score in the range of 0 (no disease) to 72 (maximal disease)
Time Frame: 4 weeks, 8 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Enstilar® Foam | Vehicle Foam
Number analyzed (Participants) | 19 | 5
Participants
  4 weeks | 12 | 0
  8 weeks | 11 | 1

3. Secondary Outcome: Number of Patients Achieving Targeted Psoriasis Scalp Severity Index (PSSI)
Description: Number of patients achieving ≥50% improvement and/or ≥75% improvement in PSSI at weeks 2, 4 and 8. The Psoriasis Scalp Severity Index (PSSI) assesses severity of scalp disease along the parameters of erythema, induration, and desquamation. The PSSI uses a 5-point scale to grade the three aforementioned clinical parameters. The parameters scores are summed and multiplied by an integer (0-6) that represents the area of affected scalp. The PSSI score ranges from 0 (no disease) to 72 (maximal disease).
Time Frame: 2 weeks, 4 weeks, 8 weeks
Population: Variation in N due to # of patients who completed study visits at each timepoint.
Measure: Count of Participants; unit: Participants
Arm/Group | Enstilar® Foam | Vehicle Foam
Number analyzed (Participants) | 19 | 5
Participants
  2 weeks: number analyzed (Participants) | 19 | 3
  2 weeks | 7 | 1
  4 weeks: number analyzed (Participants) | 19 | 4
  4 weeks | 8 | 1
  8 weeks: number analyzed (Participants) | 19 | 3
  8 weeks | 9 | 2

4. Secondary Outcome: Number of Patients With Treatment Success According to Investigator Global Assessment (IGA Mod 2011)
Description: Number of patients at week 8 who achieved treatment success according to IGA mod 2011 of the entire body including scalp. IGA ranges from 0 (clear) to 4 (severe). Treatment success is defined as IGA of clear (0) or almost clear (1) for patients with ≥ moderate disease at baseline or IGA of clear (0) for patients with mild disease at baseline.
Time Frame: at week 8
Measure: Count of Participants; unit: Participants
Arm/Group | Enstilar® Foam | Vehicle Foam
Number analyzed (Participants) | 19 | 5
Participants | 3 | 0

5. Secondary Outcome: Number of Participants Who Achieved Treatment Success According to Scalp Investigator Global Assessment (ScIGA)
Description: Number of patients at weeks 4 and 8 who achieved treatment success according to ScIGA. ScIGA ranges from 0 (clear) to 4 (severe). Treatment success is defined as ScIGA of clear (0) or almost clear (1) for patients with ≥ moderate disease at baseline or ScIGA of clear (0) for patients with mild disease at baseline.
Time Frame: 4 weeks, 8 weeks
Population: Data for participants with scalp disease who completed the respective study visits.
Measure: Count of Participants; unit: Participants
Arm/Group | Enstilar® Foam | Vehicle Foam
Number analyzed (Participants) | 11 | 4
Participants
  4 weeks | 6 | 0
  8 weeks | 2 | 1

6. Secondary Outcome: Patient's Global Assessment of Itch
Description: Patient's Global Assessment of Itch as compared to baseline measured by Visual Analog Scale (VAS). The VAS is a numerical scale used to assess patients' perception of pruritus/itch.The evaluation is a 10cm long line on which the subjects indicate the severity of their pruritus from "0" (no pruritus) to "10" (severe pruritus).
Time Frame: Baseline, 2 weeks, 4 weeks, 8 weeks
Population: data only for participants who completed respective study visits
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Enstilar® Foam | Vehicle Foam
Number analyzed (Participants) | 19 | 5
score on a scale
  baseline | 6.9 (2.4) | 6.4 (2.33)
  2 weeks: number analyzed (Participants) | 19 | 3
  2 weeks | 3.6 (2.2) | 1.3 (2.3)
  4 weeks | 3.1 (2.5) | 3.2 (2.3)
  8 weeks | 2.6 (2.2) | 2.8 (1.5)

7. Secondary Outcome: Number of Participants Who Clear or Almost Clear Disease According to the Patient's Global Assessment of Disease Severity (PaGA)
Description: PaGA have 5 distinct options ranging from (0) "Clear" to (4) "Severe." Number of participants with treatment response defined as clear or almost clear disease (for those with moderate or severe disease at baseline) or clear disease (for those with mild disease at baseline) at 4 weeks and 8 weeks.
Time Frame: 4 weeks, 8 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Enstilar® Foam | Vehicle Foam
Number analyzed (Participants) | 19 | 5
Participants
  4 weeks | 6 | 1
  8 weeks | 6 | 1

8. Secondary Outcome: Erythema Indices of Target Psoriasis Plaque
Description: A skin spectrophotometer (Mexameter) was used to quantify the degree of erythema of lesional skin compared to an index area (of unaffected skin). The mexameter measures from 0-999. The higher the value for erythema index the more red pigmentation in the skin, this is assessed by quantification of hemoglobin in the skin via reflectance spectroscopy.
Time Frame: Baseline, 2 weeks, 4 weeks, 8 weeks
Population: data results for participants who completed respective study visits
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Enstilar® Foam | Vehicle Foam
Number analyzed (Participants) | 19 | 5
units on a scale
  baseline | 563.1 (39.0) | 559.8 (19.8)
  2 weeks: number analyzed (Participants) | 19 | 3
  2 weeks | 14.7 (25.2) | 22.3 (28.5)
  4 weeks | 13.2 (35.1) | 10.4 (16.8)
  8 weeks | 7.7 (26.5) | 22.4 (23.0)

9. Secondary Outcome: Melanin Indices of Target Psoriasis Plaque
Description: A skin spectrophotometer (Mexameter) was used to quantify the melanin index (degree of hyperpigmentation or hypopigmentation) of lesional skin compared to an index area of unaffected skin. The mexameter measures from 0-999. The higher the value for melanin index, the more brown pigment in the skin, this is assessed by quantification of melanin in the skin via reflectance spectroscopy.
Time Frame: Baseline, 2 weeks, 4 weeks, 8 weeks
Population: data results for participants who completed respective study visits
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Enstilar® Foam | Vehicle Foam
Number analyzed (Participants) | 19 | 5
units on a scale
  baseline | 578.8 (78.6) | 611 (98.3)
  2 weeks: number analyzed (Participants) | 19 | 3
  2 weeks | 14.0 (33.6) | -12.0 (16.1)
  4 weeks | 14.5 (37.0) | -11.8 (43.1)
  8 weeks | 25 (39.9) | -2.6 (36.9)

10. Secondary Outcome: Physician Dyspigmentation Visual Analog Scale (VAS)
Description: An investigator performed a visual analog scale (VAS) rating the degree of dyspigmentation of the skin. This VAS ranges from - 5 to 5 as follows: 5 severe dark brown pigmentation (darkest imaginable color), 4 dark brown pigmentation, 3 medium brown pigmentation, 2 light brown pigmentation, 1 slight dark pigmentation (barely perceptible compared to surrounding skin), 0 baseline skin pigmentation, -1 slight hypopigmentation (barely perceptible compared to surrounding skin), -2 mild hypopigmentation (light brown), -3 moderate hypopigmentation (creme-colored skin), -4 severe hypopigmentation (almost complete absence of pigment), -5 depigmentation (complete absence of pigment).
Time Frame: baseline, 4 weeks, 8 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Enstilar® Foam | Vehicle Foam
Number analyzed (Participants) | 19 | 5
score on a scale
  baseline | 1.26 (1.74) | 2 (1.26)
  4 weeks | -0.4 (2.5) | 0.2 (0.4)
  8 weeks | -0.5 (1.8) | -0.4 (1.1)

11. Secondary Outcome: Mean Change in Dermatology Life Quality Index (DLQI)
Description: DLQI full scale ranges from 0 (no effect at all on patient's life) to 30 (extremely large effect on patients' life). Mean change from Baseline in DLQI at 2, 4, and 8 weeks.
Time Frame: Baseline, 2 weeks, 4 weeks, 8 weeks
Population: data results for participants who completed respective study visits
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Enstilar® Foam | Vehicle Foam
Number analyzed (Participants) | 19 | 5
score on a scale
  baseline | 11.9 (5.9) | 14.4 (8.7)
  2 weeks: number analyzed (Participants) | 19 | 3
  2 weeks | -4.4 (5.3) | -11.3 (4.7)
  4 weeks | -6.5 (3.4) | -6.8 (8.7)
  8 weeks | -6.4 (5.5) | -7.2 (6.6)

ADVERSE EVENTS:
Time Frame: 8 weeks
Arm/Group | Enstilar® Foam | Vehicle Foam
All-Cause Mortality (participants affected / at risk) | 0/20 | 0/5
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/5
Other Adverse Events (participants affected / at risk) | 5/20 | 1/5
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Enstilar® Foam (N=20) | Vehicle Foam (N=5)
Common Cold (Respiratory, thoracic and mediastinal disorders) | 3 | 0
Upper Respiratory Infection (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Bee Sting (Injury, poisoning and procedural complications) | 1 | 0
Diarrhea (Gastrointestinal disorders) | 2 | 0
Upper Extremity Pain (Musculoskeletal and connective tissue disorders) | 2 | 0
Headache (General disorders) | 1 | 0
Seasonal Allergies (General disorders) | 1 | 0
Seborrheic Dermatitis (Skin and subcutaneous tissue disorders) | 1 | 0
Worsening Intertrigo (Skin and subcutaneous tissue disorders) | 1 | 0
Daytime Sleepiness (General disorders) | 1 | 0
Hypopigmented Macules (Skin and subcutaneous tissue disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2017-08-10): https://cdn.clinicaltrials.gov/large-docs/77/NCT03506477/Prot_000.pdf
  • Statistical Analysis Plan (2017-08-10): https://cdn.clinicaltrials.gov/large-docs/77/NCT03506477/SAP_001.pdf